CLINICAL TRIAL: NCT01200849
Title: Enhanced Spanish Drug Label Design to Promote Patient Understanding and Use
Brief Title: Enhanced Spanish Drug Label Study to Promote Patient Understanding and Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael S. Wolf, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00005495
Record Dates: First submitted 2010-09-02; First posted 2010-09-14 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Medication Understanding; Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Label (Experimental): Subjects in this arm will receive their prescriptions labeled with our enhanced, patient-friendly label.
  Interventions: Other: Enhanced Label
- Standard Label (No Intervention): Subjects in this arm will receive their prescriptions labeled with a standard label.

INTERVENTIONS:
Other: Enhanced Label — A prescription drug label that has simplified text, more white space and overall is more patient-friendly.
  Arms: Enhanced Label

SUMMARY:
The overall objective of this study is to test the efficacy of an evidence-based, enhanced Rx container label design to improve Spanish speaking patients' understanding of instructions for use.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial (N=960) to evaluate the efficacy of the enhanced Rx container label to improve, Spanish speaking, diabetic and/or hypertensive patients' understanding of actual prescribed medicines, compared to a standard label format. Spanish-speaking patients with type II diabetes and/or hypertension at safety-net clinics affiliated with one central-fill pharmacy (Nova Scripts Central - NSC) receive all their prescribed medicines from this location. Recruited diabetic and/or hypertensive subjects in this study will be randomly assigned to either intervention (enhanced Rx container label) or control (standard Rx label). All pill-form, regular dosing schedule medicines, including diabetes and hypertensive (i.e. ACE inhibitor) medicines associated with patients' treatment will be labeled according to study arm by the central-fill pharmacy. Study subjects will be interviewed at the time of dispensing the prescribed medicines at the clinic, again three months later (dispensing of refill), and finally nine months after baseline (dispensing of refill). Pharmacy refill data and medical record information - linked at these clinics - will be collected for exploratory analyses. Patients' ability to read and demonstrate Rx label instructions, including auxiliary warnings, will be the primary outcomes for this aim. Data from the actual use trial will be processed, reviewed, analyzed (in order of hypotheses), and reports prepared during the final months of this last phase of the study. We anticipate several manuscripts to be developed as a result of this project, supported by the diverse key personnel and collaborating faculty enlisted.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type II diabetes or hypertension in their medical chart
* Spanish speaking
* 30 years or older

Exclusion Criteria:

* Uncorrectable hearing or visual impairment.
* Too ill to participate

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Understanding of prescription medication | Baseline, 3 month follow-up, 9 month follow-up
  Difference in understanding and comprehension of medication use as compared to control.

SECONDARY OUTCOMES:
Change in HbA1c or blood pressure readings | Baseline, 3 month follow-up, 9 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolf, Phd, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Wolf MS, Davis TC, Curtis LM, Bailey SC, Knox JP, Bergeron A, Abbet M, Shrank WH, Parker RM, Wood AJ. A Patient-Centered Prescription Drug Label to Promote Appropriate Medication Use and Adherence. J Gen Intern Med. 2016 Dec;31(12):1482-1489. doi: 10.1007/s11606-016-3816-x. Epub 2016 Aug 19. PMID 27542666